CLINICAL TRIAL: NCT01465919
Title: Phase 4 Open-labeled Study to Compare the Anti-depressive Efficacy Between Mirtazapine and Psychotherapy for Patients With Interferon-related Depression During Antiviral Therapy for Hepatitis C
Brief Title: Efficacy Study of Mirtazapine to Treat Interferon-related Depression During Antiviral Therapy for Hepatitis C
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the recent change in standard of care for hepatitis C.
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Won Kim, Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-2011-130
Record Dates: First submitted 2011-10-31; First posted 2011-11-07 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Depression
Keywords: depression; interferon; chronic hepatitis C; mirtazapine
MeSH Terms: conditions — Depression; Hepatitis C, Chronic | interventions — Mirtazapine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mirtazapine (Experimental): mirtazapine
  Interventions: Drug: Mirtazapine
- Supportive psychotherapy (Other): Supportive psychotherapy will be given by a specialized psychiatrist.
  Interventions: Other: Supportive psychotherapy

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine will be administered at baseline, 1-week, 2-week, 4-week, 6-week, and 8-week, dosing between 7.5mg/day and 45mg/day, in patients with interferon induced depression.
  Other Names: Remeron
  Arms: mirtazapine
Other: Supportive psychotherapy — Supportive psychotherapy will be administered at baseline, 1-week, 2-week, 4-week, 6-week, and 8-week in patients with interferon induced depression.
  Other Names: psychotherapy
  Arms: Supportive psychotherapy

SUMMARY:
The purpose of this study is to evaluate the anti-depressive efficacy of mirtazapine in depression induced by peginterferon alpha-2a and ribavirin treatment in Korean patients with chronic hepatitis C.

DETAILED DESCRIPTION:
Depression is a common serious adverse event (30%-50%) during the interferon treatment for chronic hepatitis C. Adequate control of depressive symptoms might enable to adhere to antiviral therapy and lead to the favorable prognosis for patients with chronic hepatitis C.

Mirtazapine is an effective antidepressant for depressive mood as well as insomnia and anxiety. Mirtazapine has also relatively lower drug-drug interactions, which are important for patients with hepatic dysfunction.

In this study, the investigators are going to perform an 8-week, randomized, open label trial comparing anti-depressive efficacy between mirtazapine and supportive psychotherapy in depression induced by peginterferon alpha-2a and ribavirin treatment in Korean patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode diagnosed with Diagnostic and Statistical Manual Diploma in Social Medicine-IV (DSM-IV)
* Hamilton Depression Scale (HAMD-17) ≥ 14

Exclusion Criteria:

* Any other axis I primary diagnoses except major depressive disorder
* Having serious adverse events or hypersensitivity to mirtazapine
* Having major depressive disorder prior to the first injection of interferon

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale (HAMD)-17 at 8 weeks | Baseline and 8-week of andi-depressive treatment
  depression change

SECONDARY OUTCOMES:
Change from baseline in quality of life at 8 weeks | Baseline and 8-week of andi-depressive treatment
  Psychometric assessment of quality of life using The Brief Form of the World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) and Liver Disease Quality of Life (LDQOL)
Genetic polymorphism | Baseline
  Determination of genetic factors (single nucleotide polymorphism) as predictors of clinical responses to mirtazapine in interferon-induced depression.

CONTACTS AND LOCATIONS:
Overall Officials: Won Kim, MD, PhD, Principal Investigator — Seoul Metropolitan Government Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi JS, Kim W, Sohn BK, Lee JY, Jung HY, Oh S, Joo SK, Kim HY, Jung YJ. Association of Changes in Mood Status and Psychosocial Well-Being with Depression During Interferon-Based Treatment for Hepatitis C. Psychiatry Investig. 2017 May;14(3):314-324. doi: 10.4306/pi.2017.14.3.314. Epub 2017 May 16. PMID 28539950